CLINICAL TRIAL: NCT06232863
Title: A Phase I Study To Evaluate The Safety, Tolerability and Pharmacokinetics Of BH009 In Patients With Advanced Head And Neck Squamous (Non-nasopharyngeal) And Ovarian Cancer
Brief Title: A Study of BH009 in Head and Neck Squamous Cell Carcinoma and Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuhai Beihai Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH009-I-101; CTR20230004 (Other: NMPA)
Record Dates: First submitted 2024-01-19; First posted 2024-01-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult
Keywords: Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BH009 (Experimental): Every 28 days constitutes a treatment cycle, and administration on day 1, day 8, day 15 of each cycle
  Interventions: Drug: BH009

INTERVENTIONS:
Drug: BH009 — Every 28 days constitutes a treatment cycle, and administration on day 1, day 8, day 15 of each cycle

SUMMARY:
This study will assess the safety and tolerability and pharmacokinetics of BH009 in patients with advanced head and neck squamous (non-nasopharyngeal) and ovarian cancer.

DETAILED DESCRIPTION:
This is a multicenter, open label phase I clinical study to evaluate the safety, tolerability, and pharmacokinetic profile of BH009 in patients with advanced squamous head and neck cancer (non-nasopharyngeal) and ovarian cancer, and to initially explore its clinical effectiveness. This study will use a "3+3" dose escalation design to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of BH009.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18-70 years old at the time of informed consent.
2. Histologically or cytologically proven squamous cell carcinoma of the head and neck(including oropharynx, oral cavity, hypopharynx and larynx, excluding nasopharyngeal carcinoma) and ovarian carcinoma (including epithelial ovarian carcinoma, fallopian tube carcinoma and primary peritoneal carcinoma).
3. Subjects who failed by standard treatments, or refused standard treatments, or the investigator considered the subject unsuitable for standard treatments.
4. At least one measurable lesion according to RECIST 1.1 at baseline.
5. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Subjects must have an expected survival of at least 3 months.
7. Subjects must have adequate organ and marrow function. Laboratory results meet the following conditions within 7 days prior to the first dose [subjects must not have received recombinant granulocyte-colony stimulating factor (G-CSF) or blood transfusion within 14 days prior to the first dose]:

   * Hematological : Absolute neutrophil count(ANC)≥1.5×109/L, platelet count(PLT)≥100×109/L, hemoglobin(Hb)≥90 g/L;
   * Renal function :Serum creatinine(Cr)≤1.5×ULN and creatinine Clearance ≥50 mL/min(Cockcroft-Gault );
   * Liver function : Total bilirubin ≤1.5×ULN, alanine aminotransferase(ALT)and aspartate aminotransferase(AST) ≤ 1.5×ULN (if liver tumor/metastases are present, then ≤2.5×ULN is allowed).
8. Subjects with a left ventricular ejection fraction of ≥50% measured by echocardiography at baseline, a normal 12-lead electrocardiogram or no clinically significant abnormalities, QTc intervals <450 ms (men) or <470 ms (women) (Fridericia's), and no signs or symptoms of heart failure.
9. Subjects with remission of toxicity due to prior therapy to ≤ grade 1 (except for toxicities such as alopecia that are not considered a safety risk by investigator).
10. Subjects have not received surgery, chemotherapy, radiotherapy, immunotherapy, biotherapy, targeted therapy, anti-tumour herbs, small molecule targeted drugs, within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of the drug.
11. Subjects voluntarily signed the informed consent form, had good compliance, were available for follow-up, and voluntarily complied with study regulations.

Exclusion Criteria:

1. Subjects with a known hypersensitivity to the study drug and any excipient contained in the drug formulation,or intolerance to paclitaxel analogues.
2. Subjects are currently receiving other anti-tumor therapy.
3. Subjects requiring a potent inhibitor of CYP3A4 within 14 days prior to the first dose and during the study period.
4. Subjects have been treated with systemically administered glucocorticosteroid (prednisone > 10 mg/day or equivalent dose of other similar drug) or other immunosuppressive agents within 14 days prior to the first use of the investigational medicinal product; with the exception of the following: treatment with topical, ophthalmic, intra-articular, intranasal, and inhaled glucocorticosteroids; and short-term prophylactic glucocorticosteroids (e.g., prevention of allergy to contrast media).
5. Subjects with clinically significant psychiatric or central nervous system disorders.
6. Subjects with a primary malignant tumour of the brain; or those who with two or more malignant tumours (except cured non-melanoma skin cancer, cervical cancer, thyroid cancer and intramucosal cancer of the gastrointestinal tract).
7. Subjects who with serious medical conditions:

   * Subjects with clinically significant cardiovascular disease, including: severe or uncontrolled heart disease requiring treatment, congestive heart failure classified by the New York Heart Association (NYHA) as grade 3 or 4, unstable angina pectoris uncontrolled by medication, history of myocardial infarction within 6 months prior to enrolment, severe arrhythmia requiring medication (except atrial fibrillation or paroxysmal supraventricular tachycardia);
   * Subjects with indwelling cardiac stents within 6 months;
   * Subjects with uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg after pharmacological intervention), diabetes mellitus (glycated haemoglobin HbA1c ≥8.0% or fasting blood glucose ≥10.0 mmol/L), pleural effusion, pericardial effusion, ascites;
   * Subjects have uncontrolled peptic ulcer, or other uncontrolled thromboembolic event;
   * Subjects with interstitial lung disease, pulmonary fibrosis, or a history of pneumonia requiring steroid therapy.
8. Subjects with known HIV, HBV, HCV, and syphilis spirochete infections (hepatitis B surface antigen (HBsAg)-positive with HBV-DNA greater than 1,000 IU/mL; HCV-Ab-positive with a copy number higher than the upper limit of normal on the HCV RNA assay); and uncontrolled active infections (in those requiring systemic anti-infective therapy, or subjects with a temperature of >38°C (axillary temperature) prior to dosing and unable to explain it).
9. Subjects have a history of drug abuse.
10. Pregnant or nursing women; positive pregnancy test within 7 days prior to the first dose in female subjects of childbearing potential; any female subjects of childbearing potential does not consent to use of a medically recognised effective method of contraception throughout the trial period and for 3 months after the the last dose.
11. Subjects who have been participated in other clinical trial within 28 days prior to the first dose (from the date of the last dose).
12. Subjects who have been vaccinated within 28 days prior to the first dose or who will be vaccinated throughout the study (except for inactivated vaccines).
13. Subjects who be unsuitable for inclusion by investigators judgement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | first dose to 30 days after last dose
  All adverse events (AE) defined by CTCAE version 5.0
Recommended phase 2 dose of BH009 | first dose to 30 days after last dose
  defined by CTCAE version 5.0
MTD of BH009 | first dose to 30 days after last dose
  When the dose is incremented beyond the MTD, the previous lower dose group will be identified as the MTD.

SECONDARY OUTCOMES:
Objective response rate | After first dose until 30 days after last dose
  Objective response rate by RECIST version 1.1
Duration of relief | After first dose until 30 days after last dose
  Duration of relief by RECIST version 1.1
Disease control rate | After first dose until 30 days after last dose
  Disease control rate by RECIST version 1.1
Progression-free survival | After first dose until 30 days after last dose
  Disease control rate by RECIST version 1.1
PK Analysis of BH009 | predose, 30 minutes, 45 minutes, 1 hour after the start of infusion (immediately after the end of infusion), 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after the end of infusion
  Maximum Concentration (Cmax)
PK Analysis of BH009 | predose, 30 minutes, 45 minutes, 1 hour after the start of infusion (immediately after the end of infusion), 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after the end of infusion
  Time to Cmax (Tmax)
PK Analysis of BH009 | predose, 30 minutes, 45 minutes, 1 hour after the start of infusion (immediately after the end of infusion), 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after the end of infusion
  Area Under the Curve From Time 0 Hours to Last Quantifiable Concentration (AUC0-last)
PK Analysis of BH009 | predose, 30 minutes, 45 minutes, 1 hour after the start of infusion (immediately after the end of infusion), 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after the end of infusion
  Area Under the Curve From Time 0 Hours to Infinity (AUC0-inf)
PK Analysis of BH009 | predose, 30 minutes, 45 minutes, 1 hour after the start of infusion (immediately after the end of infusion), 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after the end of infusion
  Apparent Terminal Elimination Half-Life (t1/2)
PK Analysis of BH009 | predose, 30 minutes, 45 minutes, 1 hour after the start of infusion (immediately after the end of infusion), 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after the end of infusion
  Apparent Total Clearance (CL)
PK Analysis of BH009 | predose, 30 minutes, 45 minutes, 1 hour after the start of infusion (immediately after the end of infusion), 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after the end of infusion
  Apparent Volume of Distribution (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, PI, Principal Investigator — Hunan Cancer Hospital; Yaqian Han, PI, Principal Investigator — Hunan Cancer Hospital
Locations (5):
- China (5):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affiliated Zhongshan Hospital Of Dalian University, Dalian, Liaoning
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No